CLINICAL TRIAL: NCT06593522
Title: A Phase 2 Study Evaluating the Efficacy, Safety, Tolerability, and Pharmacokinetics of AMG 193 in Subjects With Methylthioadenosine Phosphorylase (MTAP)-Deleted Previously Treated Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Phase 2 Study of AMG 193 in Participants With MTAP-deleted Advanced NSCLC (MTAPESTRY 201)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20230153
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: MTAP-deleted NSCLC
Keywords: Oncology; AMG 193
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Evaluation (Experimental): Participants will be randomized to receive one of 2 active dose levels of AMG 193 orally (PO) daily (QD) in 28 days cycles. Part 1 of the study will determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: AMG 193
- Part 2: Dose Expansion (Experimental): Participants will receive AMG 193 PO QD in 28-day cycles at the RP2D.
  Interventions: Drug: AMG 193

INTERVENTIONS:
Drug: AMG 193 — Film-coated tablet

SUMMARY:
The main objective of the study is to characterize safety and efficacy of 2 dose levels of AMG 193 by investigator, and to evaluate AMG 193 monotherapy efficacy by Blinded Independent Central Review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable locally advanced MTAP-deleted (Homozygous deletion of MTAP) NSCLC
* Participants will have received and progressed or experienced disease recurrence on or after receiving at least 1 prior systemic therapy for locally advanced and unresectable or metastatic disease.
* Either an archival tissue sample or an archival block must be available.
* Life expectancy of greater than 3 months, in the opinion of the investigator.
* Participants who have had brain metastases and have been appropriately treated with radiation therapy or surgery ending at least 14 days before study day 1 are eligible.
* Participants with untreated asymptomatic brain metastases smaller or equal to 2 cm in size (per lesion if more than one) and not requiring corticosteroid treatment are eligible.

Exclusion Criteria:

Disease Related

• Tumors harboring the following mutations amenable to targeted therapies: epidermal growth factor receptor (EGFR), ALK receptor tyrosine kinase (ALK), ROS proto-oncogene 1 (ROS1), neurotrophic tyrosine receptor kinase (NTRK), MET proto-oncogene (MET), B-Raf proto-oncogene (BRAF), RET proto-oncogene (RET), Human epidermal growth factor receptor 2 (HER2/ERBB2), KRAS proto-oncogene G12C (KRAS G12C).

Other Medical Conditions

* Major surgery within 28 days of study day 1.
* Untreated symptomatic central nervous system (CNS) metastatic disease regardless of size or asymptomatic brain metastases greater than 2 cm per lesion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2028-11-29 (Estimated); Study Completion 2030-11-29 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) per RECIST 1.1 | Up to 35 months
Objective response (OR) Measured by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) and Assessed per Response Evaluation Criteria in Solid Tumors v1.1 (RECIST 1.1) | Up to 35 months
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to 35 months
Number of Participants Experiencing Events of Interest (EOIs) | Up to 35 months
Maximum Concentration (Cmax) of AMG 193 | Cycle 1: Day 1 and Day 15 pre-dose, 0.5 hours, 1 hour, 2 hours, 4 hours, and 6 hours post-dose; Cycle 2: Day 1 and Day 15 pre-dose; Cycles 3-5: Day 1 pre-dose
Time to Cmax (Tmax) of AMG 193 | Cycle 1: Day 1 and Day 15 pre-dose, 0.5 hours, 1 hour, 2 hours, 4 hours, and 6 hours post-dose; Cycle 2: Day 1 and Day 15 pre-dose; Cycles 3-5: Day 1 pre-dose
Area Under The Concentration-time Curve (AUC) of AMG 193 | Cycle 1: Day 1 and Day 15 pre-dose, 0.5 hours, 1 hour, 2 hours, 4 hours, and 6 hours post-dose; Cycle 2: Day 1 and Day 15 pre-dose; Cycles 3-5: Day 1 pre-dose

SECONDARY OUTCOMES:
Disease Control (DC) by BICR | Up to 35 months
Duration of Response (DOR) by BICR | Up to 35 months
Time to Response (TTR) by BICR | Up to 35 months
Progression-free Survival (PFS) by BICR | Up to 35 months
OR by Investigator's Assessment | Up to 35 months
DC by Investigator's Assessment | Up to 35 months
DOR by Investigator's Assessment | Up to 35 months
TTR by Investigator's Assessment | Up to 35 months
PFS by Investigator's Assessment | Up to 35 months
Overall Survival (OS) | Up to 35 months
Number of Participants Experiencing TEAEs | Up to 35 months
Cmax of AMG 193 | Cycle 1: Day 1 and Day 15 pre-dose, 0.5 hours, 1 hour, 2 hours, 4 hours, and 6 hours post-dose; Cycle 2: Day 1 and Day 15 pre-dose; Cycles 3-5: Day 1 pre-dose
Tmax of AMG 193 | Cycle 1: Day 1 and Day 15 pre-dose, 0.5 hours, 1 hour, 2 hours, 4 hours, and 6 hours post-dose; Cycle 2: Day 1 and Day 15 pre-dose; Cycles 3-5: Day 1 pre-dose
AUC of AMG 193 | Cycle 1: Day 1 and Day 15 pre-dose, 0.5 hours, 1 hour, 2 hours, 4 hours, and 6 hours post-dose; Cycle 2: Day 1 and Day 15 pre-dose; Cycles 3-5: Day 1 pre-dose
Change in Quality of life (QoL) per The European Organization for Research and Treatment of Cancer Quality of life Questionnaire (EORTC QLQ)-C30 | Up to 12 months
Change in QoL per Quality of Life Questionnaire-Lung Cancer 13 (QLQ LC13) | Up to 12 months
Change in QoL per European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) | Up to 12 months
Overall Health Status per Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 12 months
Overall Health Status per The Functional Assessment of Cancer Therapy - General (FACT-G) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (91):
- United States (20):
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Hartford HealthCare Cancer Institute - Manchester, Plainville, Connecticut
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Our Lady of the Lake Cancer Institute, Baton Rouge, Louisiana
  - Trinity Health Saint Joseph Mercy Ann Arbor, Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - Texas Oncology Central/South Texas, Austin, Texas
  - Sarah Cannon Research Institute, Dallas, Texas
  - Texas Oncology - Dallas Fort Worth, Dallas, Texas
  - US Oncology Research Investigational Products Center, Irving, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists PC, Fairfax, Virginia
- Australia (4):
  - GenesisCare -North Shore Oncology, St Leonards, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
- Brazil (10):
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Fundacao pio xII Barretos, Barretos, São Paulo
  - Fund Faculdade Regional Med Sao Jose Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer Estado SP Icesp, São Paulo, São Paulo
  - Fundacao Antonio Prudente - Hosp AC Camargo, São Paulo, São Paulo
  - Instituto de Educacao Pesquisa e Gestao em Saude, Rio de Janeiro
  - Centro Paulista de Oncologia, São Paulo
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - William Osler Health System - Brampton Civic Hospital, Brampton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre Glen Site, Montreal, Quebec
- China (14):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni Thomayerova nemocnice, Prague
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Japan (6):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Netherlands (3):
  - Nederlands Kanker Instituut Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - Sint Jansdal Ziekenhuis, Harderwijk
  - Erasmus Medisch Centrum, Rotterdam
- Portugal (4):
  - Unidade Local de Saude de Braga, EPE, Braga
  - Fundacao Champalimaud, Lisbon
  - Hospital Cuf porto, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (4):
  - Cha Bundang Medical Center, Cha University, Seongnam-si, Gyeonggi-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon-si Gyeonggi-do
  - The Catholic University of Korea St Vincents Hospital, Suwon-si, Gyeonggi-do
- Switzerland (3):
  - Universitaetsspital Basel, Basel
  - Hopitaux Universitaires de Geneve, Geneva
  - Kantonsspital Sankt Gallen, Sankt Gallen
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Memorial Bahcelievler Hastanesi, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com